CLINICAL TRIAL: NCT04788810
Title: Toxicokinetic Study of Dichlorobisphenol A After an Oral or Dermal Single Dose in Healthy Volunteer.
Acronym: PRECEPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A02116-33
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetic Study
Keywords: Toxicokinetics; Endocrine Disruptors; Bisphenol A derivatives

STUDY DESIGN:
Intervention Model Description: Oral route = 6 volunteers Dermal route = 6 volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral route (Experimental): Volunteers receiving d12-Cl2BPA via oral route
  Interventions: Other: Administration of d12-Cl2BPA
- Dermal route (Experimental): Volunteers receiving d12-Cl2BPA via oral route
  Interventions: Other: Administration of d12-Cl2BPA

INTERVENTIONS:
Other: Administration of d12-Cl2BPA — Administration of d12-Cl2BPA

SUMMARY:
The objective of this study is to determine toxicokinetic parameters of deuterated d12-Cl2BPA after the administration of a single low dose (50 µg/kg) to healthy volunteers via oral or dermal routes.

DETAILED DESCRIPTION:
Dichlorobisphenol A (Cl2BPA)is formed by the reaction of chlorine with bisphenol A present in water during water disinfection process. As a consequence, Cl2BPA is present in various aqueous media including tap water. Cl2BPA has also been found in human, in blood, urine, breast milk and adipose tissue suggesting chronic exposure to this compound. Cl2BPA is an endocrine disruptor that binds to estrogenic and PPAR-γ receptors. Epidemiological studies have shown that exposure to DCBPA has been related to the occurrence of diabetes, obesity and myocardial infarction.

Currently, no toxicokinetic data are available to estimate the disposition (ADME) of Cl2BPA after oral and dermal exposure in human while these data are needed for proper risk assessment of this compound.

The objective of this study is to determine toxicokinetic parameters of deuterated d12-Cl2BPA after the administration of a single low dose (50 µg/kg) to healthy volunteers via oral or dermal routes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-51 year old
* No current disease
* BMI range: 18.5-24.9 kg/m²,
* Non smoker
* Normal renal function
* Normal hepatic function
* Normal gastrointestinal function
* Affiliated to national health insurance
* Having signed an informed consent

Exclusion Criteria:

* Renal function ≤ 90 ml/min/1.73 m² (CKD-EPI)
* Altered hepatic function ASAT > 50 UI/L and/or ALAT > 50 UI/L,
* Current disease,
* Heavy alcohol consumption
* No treatment susceptible to alter Cl2BPA toxicokinetics (drugs that interact with metabolic enzymes or transporter proteins,, anti-acids, etc)
* Pregnant women, lactating mothers and women of childbearing potential with no reliable medical contraception

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Hour 0-Hour 24
  Non-compartmental and compartmental toxicokinetic analysis
Cmax | Hour 0-Hour 24
  Non-compartmental and compartmental toxicokinetic analysis
Total clearance | Hour 0 - Hour 24
  Non-compartmental and compartmental toxicokinetic analysis
Volume of distribution | Hour 0 - Hour 24
  Non-compartmental and compartmental toxicokinetic analysis

SECONDARY OUTCOMES:
Secondary toxicokinetic parameters | Hour 0 - Hour 24
  half-life

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Poitiers, Poitiers, France

REFERENCES:
- [Derived] Plattard N, Gnanasegaran R, Krekesheva A, Carato P, Dupuis A, Migeot V, Albouy M, Haddad S, Venisse N. Quantification of the Conjugated Forms of Dichlorobisphenol A (3,3'-Cl 2 BPA) in Rat and Human Plasma Using HPLC-MS/MS. Ther Drug Monit. 2023 Aug 1;45(4):554-561. doi: 10.1097/FTD.0000000000001074. Epub 2023 Jan 16. PMID 36649713